CLINICAL TRIAL: NCT07171697
Title: Mindful-Med: the Evaluation of the Mindfulness-based Stress-coping and Burnout Prevention Programme for Medical Interns.
Acronym: Mindful-Med
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mindful-Med 2025; Mindful-Med (Other: RCSI)
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Stress (Psychology); Burnout; Mindfulness
MeSH Terms: conditions — Burnout, Psychological | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: 4 week tailored mindfulness and psychoeducation programme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receipt of mindfulness programme (Other)
  Interventions: Behavioral: Mindfulness and psycho-education

INTERVENTIONS:
Behavioral: Mindfulness and psycho-education — 4 week tailored mindfulness and psychoeducation programme for medical interns

SUMMARY:
The aim of this study is to evaluate the feasibility and acceptability of a mindfulness-based healthcare education (MBHC) programme with medical interns. Specific objectives are to:

* Recruit at least 24 participants to the study.
* Examine the feasibility (recruitment and retention rates) and acceptability of the MBHC programme.
* Conduct a focus group process evaluation, exploring the interns' perceptions of the MBHC programme, including their adherence to and views on the acceptability of the MBHC programme for medical interns.

ELIGIBILITY:
Inclusion Criteria:

* Working as a medical intern within RCSI hospital

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Burnout | Up to 4 weeks
  Maslach Burnout Inventory - The Maslach Burnout Inventory (MBI) (Maslach et al., 1996) is a measure of work-related burnout (Crowder and Sears, 2017). It comprises twenty-two items, with three subscales which assess: (1) Emotional exhaustion, (2) Depersonalisation of service users, (3) Personal achievement. The scale is scored on a seven-point Likert scale (0 = never; 6 = everyday). The subscales highlight levels of burnout, with differing cut-off points specified for each subscale. The emotional exhaustion subscale ranges from low levels of burnout (seventeen or less), through moderate levels of burnout (eighteen to twenty-nine), to high levels of burnout (thirty or more). The depersonalisation of service users subscale ranges from low-level burnout (five or less), through moderate burnout (six to eleven), to high-level burnout (twelve or more).
Stress | Up to 4 weeks
  Perceived Stress Scale - The Perceived Stress Scale (PSS) (Cohen et al., 1983) is widely used to assess an individual's perception of stress. It comprised ten items developed to assess how unpredictable or uncontrollable participants feel their lives are (Cohen, 1994). The scale is scored on a five-point Likert scale (0 = never; 4 = very often), with higher scores indicative of greater levels of stress.

SECONDARY OUTCOMES:
Mindfulness | Up to 4 weeks
  Southampton Mindfulness Questionnaire - The Southampton Mindfulness Questionnaire (SMQ) (Chadwick et al., 2008) is a measure which assesses aspects of individual mindfulness resulting from unpleasant thoughts and images comprising of sixteen items. It is scored on a seven-point Likert scale (0 = Disagree totally; 6 = Agree totally), with higher scores indicative of greater mindfulness. The scale comprises four, four-item, subscales assessing (i) Mindful observation (SMQ-MO); (ii) Non-attachment (SMQ-NA); (iii) Aversion (SMQ-Av); (iv) Non-judgement (SMQ-NJ).

CONTACTS AND LOCATIONS:
Locations (1):
- Alan Maddock, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No